CLINICAL TRIAL: NCT01993303
Title: Direct Comparison of 2D Cardiac PET With 3D Cardiac PET Using a 3D Monte-Carlo Scatter COrrection Algorithm
Brief Title: Direct Comparison of 2D Cardiac PET With 3D Cardiac PET
Status: Completed | Type: Observational
Sponsor: Cardiovascular Imaging Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: CVIT-01-2012
Record Dates: First submitted 2012-08-01; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Perfusion Imaging; PET; Rb-82
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Cohort: Population: 19 subjects, mean age 65 years, mean BMI 30 kg/m2, 79% male. Radionuclide Dosage: Rb-82 doses were rest 53+/-5 mCi and stress 53+/-6 mCi All were stress with Dipyridamole.

SUMMARY:
Lowering the per-infusion dose of Rb-82 offers advantages of lessening radiation exposure and extending useable generator life. Prior studies have not shown equivalence of 3D vs 2D Rb-82 PET. The investigators therefore compare 3D PET after a lower Rb-82 dose (~20 mCi) processed using a Monte-Carlo driven scatter correction algorithm against conventional higher dosage (~50 mCi) 2D Rb-82 PET MPI.

DETAILED DESCRIPTION:
This study re-examines 2D an 3D myocardial perfusion PET data from 19 subjects, mean age 65 years, mean BMI 30 kg/m2, 79% male. Rest and stress scans were acquired on a Siemens Accel™ PET scanner in 2D (septa extended) and 3D (septa retracted) modes. Rb-82 doses were rest 53+/-5 mCi and stress 53+/-6 mCi. Imaging times were 2D emission scan for 3 mins (90 sec delay post Rb-82 infusion), followed by a 3 minute, 3D gated emission scan (180 sec delay). Decay and shorter acquisition times led to a 62% reduction in the effective dosage 2D vs 3D datasets. 3D images were first pre-processed using a Monte-Carlo scatter and prompt gamma correction algorithm (Imagen3D™) then reconstructed using ImagenProTM (CVIT, Kansas City, MO). Reconstructed images were evaluated using relative, 17 segment raw scores (Cedars QPET). Studies were read by consensus of 2-blinded readers for: image quality (1-4, poor-excellent), interpretive certainty (1-3, low-high) and rest perfusion using a 17 segment model (0=normal; 1-3 = mild, moderate, or severe perfusion defects). Stress segmental scores were not evaluated due to differences in imaging start time post dipyridamole infusion.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years of Age
* Have ability to provide informed consent
* Have a technically adequate rest/stress Rb-82 perfsion PET study within the past 60 days

Exclusion Criteria:

* Pregnant or nursing feamle
* Weight > 275 lbs
* Have contraindications to adenosine stress testing
* Unstable cardiac rhythm (atrial fibrillation, frequent PVCs
* PTCA or CABG within the last 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 19 subjects, mean age 65 years, mean BMI 30 kg/m2, 79% male.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2004-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quantitative Accuracy | 1 day
  To establish the quantitative accuracy of reconstructed volumes using Imagen3DTM when compared to other methods.
Visual Assessment | 1 day
  To establish that visual assessments of image quality and reader confidence using 3D data are equivalent to the other methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Lukes Hospital, Kansas City, Missouri, United States